CLINICAL TRIAL: NCT07004426
Title: Assessment of Symptomatic and Incidental Detection of Renal Cell Carcinoma Using Standard Imaging Modalities
Brief Title: Symptomatic and Incidental RCC Detection
Acronym: KIDCaD
Status: Not yet recruiting | Type: Observational
Sponsor: Charles University, Czech Republic (Other)
Collaborators: University Hospital Kralovske Vinohrady (Unknown)
Responsible Party: Sponsor
Other Study IDs: KIDCaD
Record Dates: First submitted 2025-05-27; First posted 2025-06-04 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-05

CONDITIONS: Renal Cell Carcinoma (Kidney Cancer); Benign Renal Neoplasm; Renal Carcinoma
Keywords: Renal cell carcinoma; Detection; Imaging modalities; Non-neoplastic renal lesions
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- A single patient group undergoing intervention for renal lesions
  Interventions: Procedure: Surgical treatment of renal lesions

INTERVENTIONS:
Procedure: Surgical treatment of renal lesions — Surgical treatment of renal lesions

SUMMARY:
Evaluation of the frequency of symptomatic and incidental detection of renal carcinoma at different stages depending on the imaging modality used

DETAILED DESCRIPTION:
In the Czech Republic, there is no screening program for renal cell carcinoma. Existing evidence suggests that incidental detection of this cancer tends to occur in its early stages, which are more manageable due to effective treatment options, ultimately reducing renal cancer mortality. This highlights the potential value of evaluating current imaging modalities and determining their role in secondary prevention. This cross-sectional study, based on hospital data, aims to contribute to a better understanding of this issue and to assess the effectiveness of imaging techniques in the early detection of renal cell carcinoma. Furthermore, data analysis may reveal the influence of risk factors on the detection of tumors at various stages.

ELIGIBILITY:
Inclusion Criteria:

* patients over 18 years of age undergoing surgical treatment for renal lesions

Exclusion Criteria:

* patients undergoing surgery for non-renal and urotelial carcinoma, including unknown
* patients with recurrent renal lesions

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated for renal lesions at the Urology Department of University Hospital Královské Vinohrady
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-15 (Estimated)

PRIMARY OUTCOMES:
Detection-specific renal cell carcinoma (RCC) proportions | From 2011 to 2020
  Detection-specific renal cell carcinoma (RCC) proportions, defined as the proportion of each detection type relative to all RCC cases. Results will be stratified by stage, histological type, and imaging modality.

SECONDARY OUTCOMES:
Proportion of RCC among neoplastic and non-neoplastic renal lesions | From 2011 to 2020
  Proportion of RCC among neoplastic and non-neoplastic renal lesions, stratified by investigated covariates (e.g., age, sex, smoking status, BMI, or hypertension treatment).

CONTACTS AND LOCATIONS:
Overall Officials: Jindřich Šonský, MD, Principal Investigator — Vascular surgery, University hospital Královské Vinohrady, Prague; Alexandra Gregušová, MD, Study Chair — Vascular surgery, University hospital Královské Vinohrady, Prague; Jakub Hanych, MD, Study Chair — Vascular surgery, University hospital Královské Vinohrady, Prague; Robert Grill, assoc. prof., MD, PhD, Study Director — Vascular surgery, University hospital Královské Vinohrady, Prague; Kateřina Licková, MD, PhD, Study Chair — Vascular surgery, University hospital Královské Vinohrady, Prague; Jana Malinová, MD, PhD, Study Chair — Vascular surgery, University hospital Královské Vinohrady, Prague; Tomáš Blažek, MD, PhD, Study Chair — Ostrava University Hospital
Locations (1):
- University Hospital Královské Vinohrady, Prague, Czechia

IPD SHARING:
Plan to Share IPD: Yes
The data that support the findings of this study will be available from the principal investigators upon reasonable request.
Supporting Information: CSR
Time Frame: planned from August 2025 for a period of 5 years
Access Criteria: The data that support the findings of this study will be available from the principal investigators upon reasonable request.